CLINICAL TRIAL: NCT04543487
Title: The Effect of Therapeutic Touch on Labour Pain, Anxiety and Childbirth Attitude
Brief Title: Therapeutic Touch on Labour Pain, Anxiety and Childbirth Attitude
Acronym: touch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Sukran Ertekin Pinar, Faculty of Health Sciences, Cumhuriyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TR SIVAS01
Record Dates: First submitted 2020-08-25; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: First Pregnancy; Vaginal Delivery
Keywords: therapeutic touch; labour pain; anxiety; childbirth attitude
MeSH Terms: conditions — Labor Pain; Anxiety Disorders | interventions — Therapeutic Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control Group (Experimental): Group name
  Interventions: Other: Therapeutic touch

INTERVENTIONS:
Other: Therapeutic touch — Therapeutic touch was applied twice to the women in the intervention group in addition to routine practices. The first application was performed in the active phase of the first stage of labour, and the second was done in the second stage of labour.

SUMMARY:
Introduction: Touching ensures physical, emotional and spiritual relaxation, confidence, peace, calmness and well-being, and increases self-esteem. The aim of this study is to determine the effect of therapeutic touch on labour pain, anxiety and childbirth attitude.

Methods: The sample of this randomized controlled experimental research consisted of 80 (intervention group: 40; control group: 40) women. Data were collected using a Personal Information Form, Visual Analogue Scale, State Anxiety Inventory and Childbirth Attitudes Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Having a first pregnancy
* Not having a high-risk pregnancy
* Having no health problems with the baby or herself
* Having a single foetus
* Being about to have a vaginal delivery
* Not receiving infertility treatment
* Not having a chronic physical or psychiatric diagnosis
* Agreeing to participate in the research

Exclusion criterion

-Multiparity

Ages: 19 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Scale | 6 months
  Visual Analogue Scale
Inventory | 6 months
  State Anxiety Inventory
Questionnaire | 6 months
  Childbirth Attitudes Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Sukran Ertekin Pinar, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No